CLINICAL TRIAL: NCT03457090
Title: Extracorporeal Membrane Oxygenation and Cerebral Blood Flow Velocity Evaluated by Transcranial Doppler
Brief Title: Extracorporeal Membrane Oxygenation Evaluated by Transcranial Doppler.
Acronym: ECMO-DTC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/18/0042; 2018-A00320-55 (Other: ID-RCB)
Record Dates: First submitted 2018-02-27; First posted 2018-03-07 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
Keywords: neurologic complication, transcranial Doppler ultrasound

STUDY DESIGN:
Intervention Model Description: Patient treated with Venoarterial Extracorporeal membrane oxygenation (ECMO) Realization of transcranial doppler (TCD) of the right and left middle cerebral artery in the first 48 hours of the setting up of the ECMO with joint realization of an Trans-thoracic echocardiography (TTE) then every 24 hours until the end of the using of the ECMO and the realization of TCD and TTE during the 24 hours after removal of the ECMO.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient treated with ECMO (Experimental): Patient treated with ECMO will have Examination : a TCD and Trans-Thoracic Echocardiography (TTE)
  Interventions: Other: Examination : a TCD and Trans-Thoracic Echocardiography

INTERVENTIONS:
Other: Examination : a TCD and Trans-Thoracic Echocardiography — Examination that involves the completion of a TCD and an TTE (Trans-Thoracic Echocardiography) :
  * To reports clinical parameters at the time of the examination : ECG data: sinus rhythm, atrial or ventricular arrhythmia, state of consciousness, heart rate, O2 saturation
  * To review of pharmacological parameters at the time of the examination : presence of sedation; presence, type and dose of catecholamines.
  * To collect biological data from the day of the examination : Partial Pressure of O2, PaCO2 (partial pressure) and hematocrit
  * To collect possible additional examinations : brain scan, EEG. These are non-invasive exams that do not require patient displacement. Only the samples taken by the medical team as part of the treatment will be analyzed.
  Other Names: Examination that involves a TCD and an TTE

SUMMARY:
To determine how venoarterial extracorporeal membrane oxygenation (ECMO) affects cerebral blood flow velocity (CBFV) measured by transcranial doppler (TCD), to determine whether specific changes in cerebral blood flow velocity may be associated with neurologic injury and to determine modifications of CBFV after withdrawal of ECMO.

DETAILED DESCRIPTION:
Venoarterial Extracorporeal membrane oxygenation (ECMO) is used in adult with refractory cardiac failure as a life-saving measure. Adults treated with ECMO survived to hospital discharge in 21,8% to 65,4% of cases. Neurologic complications such as intracranial hemorrhage, anoxia and ischemia are major causes of death and long-term disability in ECMO patients (7% to 14%). Current neurological monitoring techniques are insufficient to predict which critically ill patient receiving ECMO therapy will suffer from neurologic injury. Even after a clinical suspicion of neurologic injury, diagnosis can be difficult. TCD is commonly used to monitor the CBFV of traumatic brain injury. There are no reports that evaluate CBFV of patients requiring ECMO therapy. Patient will have to do both echocardiography and TCD to evaluate cardiac output and CBFV. We will repeat these dopplers every 24 hours until ECMO withdrawal and one day after explantation.

ELIGIBILITY:
Inclusion Criteria:

* adult patient who receiving ECMO therapy

Exclusion Criteria:

* cervico-encephalic vasculopathy
* lacked an acoustic window allowing for adequate TCD examination
* stroke in medical past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow velocities evolution | 24 hours
  Cerebral blood flow velocities evolution over the time
The correlation of Cerebral blood flow velocities with the variation of the cardiac output and ECMO flow. | 24 hours
  The correlation with the variation of the cardiac output and ECMO flow.

SECONDARY OUTCOMES:
Relation between acute neurologic injury and variation of CBFV | 24 hours
  Relation between acute neurologic injury and variation of CBFV detected by TCD.
Modification of the CBFV detected by TCD after the withdrawal of the ECMO. | 24 hours
  Modification of the cerebral blood flow velocity (CBFV) detected by TCD after the withdrawal of the ECMO.
Relation between the CBFV, the NIRS, the cardiac flow and the ECMO flow. | 24 hours
  Relation between the CBFV (cerebral blood flow velocity), the Near Infrared Spectroscopy (NIRS), the cardiac flow and the ECMO flow.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny BOUNES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France